CLINICAL TRIAL: NCT05654636
Title: Evaluation of Sun's Scoring System Use in Post-pancraticodoudenectomy Pancreatic Fistula; an Observational Cohort Study.
Brief Title: Evaluation of Sun's Scoring System Use in Post-pancraticodoudenectomy Pancreatic Fistula
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Saber Mekhemer, Evaluation of Sun's scoring system use in post-pancraticodoudenectomy pancreatic fistula; an observational cohort study, Assiut University
Other Study IDs: Pancreatic fistula post PD
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Risk Scoring System for Prediction of Pancreatic Fistula Post PD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of sun scoring system for predication of pancreatic fistula after Pancreaticoduodenectomy to facilitate timely intervention after Pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is the only option curative intended in the treatment of resectable pancreatic ductal adenocarcinomas, duodenal carcinoma, ampullary carcinoma, lower common bile duct cholangiocarcinoma,. It is still associated with very high morbidity and mortality. [1]. Pancreatic cancer ranks as the seventh leading cause of cancer-related death worldwide, and the fourth among other cancers[2,3]. Pancreatic fistula(PF) is one of the most important complications after Pancreaticoduodenectomy, with an incidence of about 10% to 28%.[4].There are multiple risk factors for the predication of development of pancreatic fistula after pancreaticoduodenectomy which include soft gland texture, non-pancreatic cancer non-chronic pancreatitis pathology, small pancreatic duct diameter (<3 mm), and high intraoperative blood loss (>1000 mL) , excess intraoperative fluid administration and increased pancreatic parenchymal remnant volume [5,6,7]. Other reported risk factors as increased body mass index (BMI), poor preoperative nutrition, and male gender which preoperative may lead to pancreatic fistula [8.9]. Recent studies are deficient in evaluation and predication of pancreatic fistula . So the interest of our study to evaluate and predicate the risk factors and management of pancreatic fistula after Pancreaticoduodenectomy .

ELIGIBILITY:
Inclusion Criteria:

* All the cases indicated for Pancreaticoduedenectomy with :

  1. age less than 70 years.
  2. resectable tumour,
  3. fitness patients

Exclusion Criteria:

* 1_patients with jaundice with serum bilirubin above 200mml/dl. 2_patients with bleeding tendency until corrected. 3_patients with advanced and metastatic malignancy. 4_patients with cardiopulmonary diseases.

Ages: 25 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Assuit university hospitals which candidate for pancreaticoduodenectomy at the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
predication of pancreatic fistula after Pancreaticoduodenectomy to facilitate timely intervention after Pancreaticoduodenectomy | Baseline
  Early prediction of pancreatic fistula post PD facilities threraputic intervention and life saving in some cases

SECONDARY OUTCOMES:
Reduce the morbidity and mortality and improve the quality after pancraticoduodenectomy | Baseline
  Management of pancreatic fistula post PD improve quality of life

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Y, Zhou F, Zhu DM, Zhang ZX, Yang J, Yao J, Wei YJ, Xu YL, Li DC, Zhou J. Novel risk scoring system for prediction of pancreatic fistula after pancreaticoduodenectomy. World J Gastroenterol. 2019 Jun 7;25(21):2650-2664. doi: 10.3748/wjg.v25.i21.2650. PMID 31210716
- [Background] Chen JY, Feng J, Wang XQ, Cai SW, Dong JH, Chen YL. Risk scoring system and predictor for clinically relevant pancreatic fistula after pancreaticoduodenectomy. World J Gastroenterol. 2015 May 21;21(19):5926-33. doi: 10.3748/wjg.v21.i19.5926. PMID 26019457
- [Background] Xia W, Zhou Y, Lin Y, Yu M, Yin Z, Lu X, Hou B, Jian Z. A Predictive Risk Scoring System for Clinically Relevant Pancreatic Fistula After Pancreaticoduodenectomy. Med Sci Monit. 2018 Aug 16;24:5719-5728. doi: 10.12659/MSM.911499. PMID 30113999